CLINICAL TRIAL: NCT00919685
Title: Investigations of New Markers in Patients With Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2009/03; 2009-A00105-52
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Shock State
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: blood sample — from rest of blood sample collected for other measurements

SUMMARY:
Shock is a severe deficiency in oxygen at the cell level which could lead to the death.The study was aimed at finding markers of treatment response in patients with shock, with a better accuracy than that of lactate actually used : hypoxia-inducible factor (HIF), circulating DNA (cDNA), and plasma from cells (MPs).

DETAILED DESCRIPTION:
Shock is a severe deficiency in oxygen at the cell level which could lead to the death. The treatment strategy relies on the profile of plasma lactate level, which the kinetics and metabolism are inadequate for evaluating the treatment efficiency without delay. Hence, it is now critical to identify adequate markers of dysoxia.

The study was aimed at finding markers of treatment response in patients with shock, with a better accuracy than that of lactate.To this purpose, a multiple approach is undertaken with the analysis of 3 independent markers of cellular ischemia : hypoxia-inducible factor (HIF), circulating DNA (cDNA), and plasma from cells (MPs). Indeed, the characteristics of HIF as marker of cell dysoxia, and MPs as markers of cell apoptosis, combined with cDNA seem providing complementary information in order to describe the consequences of shock as well as the response to treatment.

Samples of patients will be collected (from rest of blood sample collected for other measurements) at each step of the management of these patients. The evolution of these markers will be compared with that of lactate plasma levels (standard of care). Subgroup analysis will be undertaken in relation with the cause of shock state (septic, cardiogenic, hemorrhagic).

ELIGIBILITY:
Inclusion Criteria:

* shock state defined by a rise of plasma lactate level (> 2 mmol/L)and/or refractory low blood pressure in the volume expansion requiring an introduction of catecholamines
* admission in intensive care < 6 hours

Exclusion Criteria:

* Pregnancy
* presumed survival lower than 48 hours
* absence of central venous way and arterial catheter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Demonstrate the superiority of at least one of 3 markers (HIF, MPs, cDNA) with regard to plasma lactate level for evaluating the treatment response in patients with shock | 2 years

SECONDARY OUTCOMES:
Improve the physiopathological knowledge of the patients with shock | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: jean GABERT, Principal Investigator — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France